CLINICAL TRIAL: NCT05818007
Title: The Effects of Hyaluronic Acid Gel on Oral Mucositis in Children Receiving Chemotherapy
Brief Title: Is Hyaluronic Acid Gel Effective on Oral Mucositis in Children Who Receiving Chemotherapy
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Yuzuncu Yil University (Other)
Responsible Party: Principal Investigator, Serap Keskin Tunc, associate professor, Yuzuncu Yil University
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: YYU-06/03.07.2019
Record Dates: First submitted 2023-04-05; First posted 2023-04-18 (Actual); Last update posted 2023-04-18 (Actual); Status verified 2023-04

CONDITIONS: Oral Mucositis
Keywords: mucositis; hyaluronic acid
MeSH Terms: conditions — Stomatitis; Mucositis | interventions — Hyaluronic Acid; Sodium Bicarbonate

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- hyaluronic acid (Experimental): The hyaluronic acid is a natural polysaccharide composed of D-glucuronic acid and N-acetyl-D-glucosamine and is synthesized as a linear polymer. The majority of the cells have a capacity to synthesize HA at a varying extent in the cell cycle.
  Interventions: Drug: Hyaluronic acid
- sodium bicarbonate (Active Comparator)
  Interventions: Drug: Sodium bicarbonate

INTERVENTIONS:
Drug: Hyaluronic acid — The main function of HA appears to be in tissue healing, by activating and modulating inflammatory responses, stimulating cellular proliferation, migration, and angiogenesis, inducing basal keratinocyte proliferation and re-epithelization by reducing collagen deposition and scarring
  Arms: hyaluronic acid
Drug: Sodium bicarbonate — sodium bicarbonate solution
  Arms: sodium bicarbonate

SUMMARY:
Oral mucositis (OM) is a common side effect of systemic chemotherapy (CT) in cancer patients. The aim of this study was to investigate the effect of hyaluronic acid (HA) gel on OM in children receiving CT.

ELIGIBILITY:
Inclusion Criteria:

* children who receive chemotherapy
* hospitalized patient

Exclusion Criteria:

- Allergy about using drugs

Ages: 3 Years to 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 40 (Actual)
Dates: Start 2022-04-01 (Actual); Primary Completion 2023-03-01 (Actual); Study Completion 2023-04-01 (Actual)

PRIMARY OUTCOMES:
World Health Organization Common Toxicity Criteria Scale | day 1st
  The lesions were classified as Grade 0 = absent; Grade 1 = pain and erythema; Grade 2 = erythema and ulcers with no difficulty in swallowing solid food; Grade 3 = ulcers requiring only liquid diet; and Grade 4 = requiring parenteral and enteral nutrition support.
World Health Organization Common Toxicity Criteria Scale | day 2nd
  The lesions were classified as Grade 0 = absent; Grade 1 = pain and erythema; Grade 2 = erythema and ulcers with no difficulty in swallowing solid food; Grade 3 = ulcers requiring only liquid diet; and Grade 4 = requiring parenteral and enteral nutrition support.
World Health Organization Common Toxicity Criteria Scale | day 3rd
  The lesions were classified as Grade 0 = absent; Grade 1 = pain and erythema; Grade 2 = erythema and ulcers with no difficulty in swallowing solid food; Grade 3 = ulcers requiring only liquid diet; and Grade 4 = requiring parenteral and enteral nutrition support.
World Health Organization Common Toxicity Criteria Scale | day 4th
  The lesions were classified as Grade 0 = absent; Grade 1 = pain and erythema; Grade 2 = erythema and ulcers with no difficulty in swallowing solid food; Grade 3 = ulcers requiring only liquid diet; and Grade 4 = requiring parenteral and enteral nutrition support.
World Health Organization Common Toxicity Criteria Scale | day 5th
  The lesions were classified as Grade 0 = absent; Grade 1 = pain and erythema; Grade 2 = erythema and ulcers with no difficulty in swallowing solid food; Grade 3 = ulcers requiring only liquid diet; and Grade 4 = requiring parenteral and enteral nutrition support.
World Health Organization Common Toxicity Criteria Scale | day 6th
  The lesions were classified as Grade 0 = absent; Grade 1 = pain and erythema; Grade 2 = erythema and ulcers with no difficulty in swallowing solid food; Grade 3 = ulcers requiring only liquid diet; and Grade 4 = requiring parenteral and enteral nutrition support.
World Health Organization Common Toxicity Criteria Scale | day 7th
  The lesions were classified as Grade 0 = absent; Grade 1 = pain and erythema; Grade 2 = erythema and ulcers with no difficulty in swallowing solid food; Grade 3 = ulcers requiring only liquid diet; and Grade 4 = requiring parenteral and enteral nutrition support.
World Health Organization Common Toxicity Criteria Scale | day 11th
  The lesions were classified as Grade 0 = absent; Grade 1 = pain and erythema; Grade 2 = erythema and ulcers with no difficulty in swallowing solid food; Grade 3 = ulcers requiring only liquid diet; and Grade 4 = requiring parenteral and enteral nutrition support.
VAS pain score | Day 1st
  A Visual Analogue Scale (VAS) is one of the pain rating scales between 1-10.
VAS pain score | Day 2nd
  A Visual Analogue Scale (VAS) is one of the pain rating scales between 1-10.
VAS pain score | Day 3rd
  A Visual Analogue Scale (VAS) is one of the pain rating scales between 1-10.
VAS pain score | Day 4th
  A Visual Analogue Scale (VAS) is one of the pain rating scales between 1-10.
VAS pain score | Day 5th
  A Visual Analogue Scale (VAS) is one of the pain rating scales between 1-10.
VAS pain score | Day 6th
  A Visual Analogue Scale (VAS) is one of the pain rating scales between 1-10.
VAS pain score | Day 7th
  A Visual Analogue Scale (VAS) is one of the pain rating scales between 1-10.
VAS pain score | Day 11th
  A Visual Analogue Scale (VAS) is one of the pain rating scales between 1-10.

CONTACTS AND LOCATIONS:
Locations (1):
- Yuzuncu Yil University, Van, Turkey (Türkiye)